CLINICAL TRIAL: NCT07377292
Title: Investigation of the Effectiveness of Core Stabilization Exercises in Patients With Rotator Cuff Tear
Brief Title: Effectiveness of Core Stabilization Exercises in Rotator Cuff Injuries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ahi Evran University Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Süleyman DALAR, Principal Investigator, Ahi Evran University Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AhievranUERH-FTR-SD-01
Record Dates: First submitted 2026-01-22; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Rotator Cuff Injury (RCI); Core Exercises Training
Keywords: Core exercise training; Rotator Cuff İnjury; Exercise
MeSH Terms: conditions — Rotator Cuff Injuries; Motor Activity

STUDY DESIGN:
Intervention Model Description: Three groups along with the exercise control group
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Core Stabilization Group (Active Comparator): Patients received conventional rehabilitation for the affected shoulder 5 days a week for 4 weeks and core stabilization exercises 3 days a week for 4 weeks.
  Interventions: Other: Core Stabilization Exercises; Other: Conventional Rehabilitation
- Classic Body Exercise Group (Active Comparator): Patients will receive conventional rehabilitation for the affected shoulder 5 days a week for 4 weeks, along with a classic trunk and abdominal strengthening program 3 days a week for 4 weeks.
  Interventions: Other: Classic Trunk and Abdominal Strengthening Program; Other: Conventional Rehabilitation
- Control Group (Placebo Comparator): Patients will receive conventional rehabilitation for the affected shoulder five days a week for four weeks.
  Interventions: Other: Conventional Rehabilitation

INTERVENTIONS:
Other: Core Stabilization Exercises — The program will be set up as a 35-minute session, including a 5-minute warm-up, three days a week for four weeks, under the supervision of a physical therapist. Before starting the exercise, the pelvis will be moved forward and backward to teach the lumbar and pelvic neutral positions by contracting and pulling the abdominal muscles to reduce lumbar lordosis. A neutral position will be established before each session, and care will be taken to maintain the neutral position throughout the exercise. The exercises consist of three levels and will be applied gradually. The exercises given at the beginning will be made more difficult individually according to the patients' progress. When the patient can maintain the exercise position for more than 5 seconds, they will move on to the next level. A deep breath will be taken before starting the exercise, and the breath will be exhaled during the movement. The contraction of the transversus abdominis muscle should continue while exhaling.
  Arms: Core Stabilization Group
Other: Classic Trunk and Abdominal Strengthening Program — The program will be set up for 3 days a week over 4 weeks, consisting of a 35-minute session including a 5-minute warm-up, supervised by a physical therapist. Classic Williams 1-2-3 and McKenzie exercises will be provided.
  Arms: Classic Body Exercise Group
Other: Conventional Rehabilitation — 1. Passive, assisted active, and active shoulder flexion, abduction, external rotation, and internal rotation exercises in the supine position
  2. Active shoulder range of motion (ROM) exercises in a sitting or standing position
  3. Shoulder flexion strengthening exercises
  4. Shoulder external rotator and internal rotator strengthening exercises
  5. Exercises to strengthen the lower, middle trapezius, and serratus anterior muscles
  6. Posterior capsule stretching exercises
  7. TENS (20 minutes)
  8. Cold pack (10 minutes)

SUMMARY:
The aim of this study is to investigate the effectiveness of core stabilization exercises added to conventional physical therapy in patients aged 40-60 with rotator cuff tears, compared to classic trunk and abdominal muscle strengthening exercises.

DETAILED DESCRIPTION:
Rotator cuff tears are classified as full-thickness and partial tears. Partial tears are a clinical condition commonly seen in the early stages but can often be treated with conservative methods. Partial tears can develop as a result of repetitive microtraumas, postural abnormalities, muscle imbalances, and deficiencies in the biomechanical chain. This condition affects not only the local shoulder muscles but also the scapulothoracic rhythm and trunk control. Recent studies have shown that shoulder function is closely related not only to local muscle strength but also to the integrity of the kinetic chain. The trunk (core) muscles are particularly critical for maintaining posture, transferring force during upper extremity movements, and stabilizing the distal segments. Inadequate trunk stabilization can lead to increased loads on the shoulder joint and elevated stress on the rotator cuff. Therefore, the aim of this thesis study is to examine the effectiveness of core stabilization exercises applied to individuals diagnosed with rotator cuff partial tears on pain, shoulder function, and clinical recovery, and to contribute scientifically to conservative rehabilitation approaches.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 40 to 60 years with a partial supraspinatus tear detected by MRI, reported by a radiologist, and confirmed by a physiatrist.
* Patients who test positive for at least two of the Jobe, Hawkins and Neer tests during the physical examination
* Patients with a visual analog scale (VAS) score between 3.5 and 7.4 millimeters (mm)

Exclusion Criteria:

* Participants do not wish to continue treatment for any reason
* Complete or massive rotator cuff tear
* Use of non-steroidal or steroidal anti-inflammatory drugs
* If they have received shoulder injections or physical therapy within the three months prior to the study
* History of acute trauma
* Presence of neurological disease
* History of surgery on the treated shoulder
* Symptomatic acromioclavicular joint arthritis
* Frozen shoulder

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 69 (Estimated)
Dates: Start 2026-02-25 (Estimated); Primary Completion 2026-12-25 (Estimated); Study Completion 2026-12-25 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | Before Treatment (Week 0), at the end of treatment (Week 3) and after treatment (Week 12)
  Pain intensity on the VAS (visual analog scale) is generally rated as "no pain" 0 points and "the most severe pain imaginable" 10 points (10 cm scale). Pain intensity scoring ranges are specified as <3 mild pain, 3-6 moderate pain, >6 severe pain.

SECONDARY OUTCOMES:
Tendon Thickness | Before Treatment (Week 0), at the end of treatment (Week 3) and after treatment (Week 12)
  The supraspinatus tendon will be evaluated using USG.
Shoulder Pain and Disability Index (SPADI) | Before Treatment (Week 0), at the end of treatment (Week 3) and after treatment (Week 12)
  The SPADI questionnaire is a measure consisting of a total of 13 questions with two subscales: pain and disability. The total score and all subscale scores are evaluated on a scale of 0-100. A high result indicates significant shoulder pain and restricted shoulder movement.
Range Of Motion (ROM) | Before Treatment (Week 0), at the end of treatment (Week 3) and after treatment (Week 12)
  Shoulder ROM is measured using a universal goniometer. Shoulder flexion, extension, abduction, internal rotation, and external rotation ranges are measured in the supine position.
Core Muscle Strength | Before Treatment (Week 0), at the end of treatment (Week 3) and after treatment (Week 12)
  Core muscle endurance will be assessed using the McGill core muscle endurance tests, which include the core flexor endurance test, core extensor endurance test, and core right and left side endurance tests. A stopwatch will be used for measurements, and scores will be recorded in seconds. Tests will be terminated when the test position deteriorates or when participants indicate they cannot continue the test.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırşehir Ahi Evran University, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No